CLINICAL TRIAL: NCT01014793
Title: Short and Long Term Efficacy of Combined Treatment in Controlling IGI-I Levels in Acromegaly
Brief Title: Short and Long Term Efficacy of Combined Cabergoline and Octreotide Treatment in Acromegalic Patients
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Priscilla Olim de Andrade MAttar, Federal University of Sao Paulo
Other Study IDs: Mattapr1
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Acromegaly
Keywords: Acromegaly resistant; combined-treatment; dopamine agonist
MeSH Terms: conditions — Acromegaly | interventions — Cabergoline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum for IGI-I, GH and prolactin measures
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Responders to cabergoline: patients with active disease under octreotide treatment received addition of increasing doses of cabergoline (1.0, 2.0 and 3.5mg/week)
  Interventions: Drug: cabergoline

INTERVENTIONS:
Drug: cabergoline — cabergoline doses were increased at 6-week intervals, starting at 1.0mg/week followed by 2.0 and 3.5mg/week. Hormonal evaluations (IGF-I, GH and PRL) started before the first dose and were repeated at 6-week intervals after each cabergoline dose and after cabergoline withdrawal
  Other Names: cabergoline-Dostinex

SUMMARY:
In acromegaly, nearly 40% of patients fail to control GH/IGF-I levels with somatostatin analogues (SA). Dopaminergic agonists (DA) are even less effective, but combination therapy with SA and DA normalizes IGF-I levels in 33-56% of patients in short-term studies. This study was designed to evaluate short and long term efficacy of cabergoline in controlling IGF-I levels in acromegalic patients receiving octreotide.

ELIGIBILITY:
Inclusion Criteria:

* Active disease, under octreotide treatment at least 9 months

Exclusion Criteria:

* Cabergoline allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nineteen acromegalic patients (Neuroendocrine Unit-UNIFESP)with active disease, resistant to octreotide were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Control of IGF-I levels | six months

SECONDARY OUTCOMES:
control IGI-I levels | six months

CONTACTS AND LOCATIONS:
Overall Officials: Julio Abucham, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rocheville M, Lange DC, Kumar U, Sasi R, Patel RC, Patel YC. Subtypes of the somatostatin receptor assemble as functional homo- and heterodimers. J Biol Chem. 2000 Mar 17;275(11):7862-9. doi: 10.1074/jbc.275.11.7862. PMID 10713101
- [Background] Holdaway IM, Rajasoorya RC, Gamble GD. Factors influencing mortality in acromegaly. J Clin Endocrinol Metab. 2004 Feb;89(2):667-74. doi: 10.1210/jc.2003-031199. PMID 14764779
- [Background] Melmed S, Colao A, Barkan A, Molitch M, Grossman AB, Kleinberg D, Clemmons D, Chanson P, Laws E, Schlechte J, Vance ML, Ho K, Giustina A; Acromegaly Consensus Group. Guidelines for acromegaly management: an update. J Clin Endocrinol Metab. 2009 May;94(5):1509-17. doi: 10.1210/jc.2008-2421. Epub 2009 Feb 10. PMID 19208732
- [Result] Cozzi R, Attanasio R, Lodrini S, Lasio G. Cabergoline addition to depot somatostatin analogues in resistant acromegalic patients: efficacy and lack of predictive value of prolactin status. Clin Endocrinol (Oxf). 2004 Aug;61(2):209-15. doi: 10.1111/j.1365-2265.2004.02082.x. PMID 15272916
- [Result] Selvarajah D, Webster J, Ross R, Newell-Price J. Effectiveness of adding dopamine agonist therapy to long-acting somatostatin analogues in the management of acromegaly. Eur J Endocrinol. 2005 Apr;152(4):569-74. doi: 10.1530/eje.1.01888. PMID 15817912
- [Result] Abs R, Verhelst J, Maiter D, Van Acker K, Nobels F, Coolens JL, Mahler C, Beckers A. Cabergoline in the treatment of acromegaly: a study in 64 patients. J Clin Endocrinol Metab. 1998 Feb;83(2):374-8. doi: 10.1210/jcem.83.2.4556. PMID 9467544
- [Result] Rocheville M, Lange DC, Kumar U, Patel SC, Patel RC, Patel YC. Receptors for dopamine and somatostatin: formation of hetero-oligomers with enhanced functional activity. Science. 2000 Apr 7;288(5463):154-7. doi: 10.1126/science.288.5463.154. PMID 10753124
- [Result] Jallad RS, Bronstein MD. Optimizing medical therapy of acromegaly: beneficial effects of cabergoline in patients uncontrolled with long-acting release octreotide. Neuroendocrinology. 2009;90(1):82-92. doi: 10.1159/000218323. Epub 2009 May 8. PMID 19439914
- [Result] Gatta B, Hau DH, Catargi B, Roger P, Tabarin A. Re-evaluation of the efficacy of the association of cabergoline to somatostatin analogues in acromegalic patients. Clin Endocrinol (Oxf). 2005 Oct;63(4):477-8. doi: 10.1111/j.1365-2265.2005.02329.x. No abstract available. PMID 16181243